CLINICAL TRIAL: NCT01124786
Title: A Phase II Randomized, Open-Label, Multicenter Study Comparing CO-1.01 With Gemcitabine as First-Line Therapy in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study Comparing CO-1.01 With Gemcitabine as First Line Therapy in Patients With Metastatic Pancreatic Adenocarcinoma (LEAP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-101-001
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: cancer; metastatic; pancreatic; pancreas; adenocarcinoma; gemcitabine; human equilibrative nucleoside transporter-1 (hENT1); CO-1.01; CO-101; CO101; Stage 4; Stage IV
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO-1.01 (Experimental)
  Interventions: Drug: CO-1.01
- gemcitabine (Active Comparator)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: CO-1.01 — 1250 mg/m2 intravenous infusion weekly for 3 weeks every 4 weeks
  Arms: CO-1.01
Drug: Gemcitabine — 1000 mg/m2 intravenous infusion weekly for 7 weeks followed by 1 week rest, then weekly for 3 weeks every 4 weeks
  Arms: gemcitabine

SUMMARY:
The purpose of this study is to determine whether CO-1.01 is safe and effective in the treatment of patients with metastatic pancreatic cancer and low hENT1 expression compared with gemcitabine.

DETAILED DESCRIPTION:
Pancreatic cancer is a very serious form of cancer. The majority of patients present with unresectable disease, and the condition is often not diagnosed until the cancer is relatively advanced. The standard first-line treatment for patients with unresectable pancreatic cancer is gemcitabine monotherapy. Unfortunately many of these patients fail to derive benefit from this treatment. No clinical or molecular marker has been established to predict benefit from gemcitabine therapy, so patients are treated empirically until evidence of disease progression or worsening performance status.

The potential for human equilibrative nucleoside transporter-1 (hENT1) expression to predict survival in gemcitabine-treated patients has been studied, and data suggest that patients with low levels of tumor cell hENT1 expression derive less benefit from gemcitabine treatment than patients with high levels of tumor cell hENT1 expression. These data support the hypothesis to be tested in this study that patients with pancreatic tumors expressing low levels of hENT1 will derive minimal benefit from gemcitabine, but will receive benefit from CO-1.01 (gemcitabine elaidate) which enters tumor cells in a hENT1-independent fashion.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic ductal adenocarcinoma (i.e., Stage 4).
* Histological/cytological confirmation of metastatic tissue (not primary tumor) by a central pathology laboratory (H&E stain) to ensure sufficient material is available for later hENT1 analysis.
* Adjuvant chemotherapy/radiotherapy ≥ 6 months prior to randomization.
* Palliative radiotherapy (if administered) ≥ 1 month prior to randomization.
* CT scan ≤30 days prior to randomization
* Performance Status (ECOG) 0 or 1.
* Estimated life expectancy ≥ 12 weeks.
* Age ≥ 18 years.
* Adequate hematological and biological function.
* Written consent on an Institutional Review Board/Institutional Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation.

Exclusion Criteria:

* Prior palliative chemotherapy for pancreatic cancer.
* Radical pancreatic resections (e.g., Whipple procedure) are not allowed < 6 months prior to randomization. Exploratory laparotomy, palliative (e.g., bypass) surgery, or other procedures (e.g., stents) are not allowed < 14 days prior to randomization. In both cases the patient must be sufficiently recovered and stable.
* Symptomatic brain metastases.
* Participation in other investigational drug clinical studies ≤ 30 days prior to randomization.
* Concomitant treatment with prohibited medications.
* History of allergy to gemcitabine or eggs.
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, uncontrolled intercurrent illness including active infection, arterial thrombosis, symptomatic pulmonary embolism).
* Any disorder that would hamper protocol compliance.
* Prior nonpancreatic malignancy treated with chemotherapy. Prior malignancies treated with surgery or radiotherapy alone must be in remission ≥ 3 years. The following prior malignancies are allowable irrespective of when they occurred: in situ carcinoma of the cervix, in situ ductal breast cancer, low-grade local bladder cancer, and nonmelanotic skin cancer.
* Females who are pregnant or breastfeeding.
* Refusal to use adequate contraception for fertile patients (females and males during the study and for 6 months after the last study treatment). Adequate forms of contraception are double-barrier methods (condoms or diaphragm with spermicidal jelly or foam); oral, depot, or injectable contraceptives; intrauterine devices; tubal ligation.
* Any other reason the investigator considers the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (21):
  - Arizona Center for Hematology Oncology, Glendale, Arizona
  - Wilshire Oncology Medical Group, Inc., Corona, California
  - White Memorial Medical Center, Los Angeles, California
  - Cancer Care Institute, Los Angeles, California
  - Newport Cancer Care Medical, Newport Beach, California
  - Hematology Oncology Associates, Oakland, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Hartford Hospital Clinical Research, Hartford, Connecticut
  - Oncology Associates of Bridgeport, Trumbull, Connecticut
  - Annapolis Oncology Center, Annapolis, Maryland
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Arena Oncology Associates, PC, Lake Success, New York
  - Bend Memorial Clinic, Bend, Oregon
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Cancer Specialists of South Texas, P.A., Corpus Christi, Texas
  - Valley Cancer Associates, Harlingen, Texas
  - South Texas Oncology and Hematology, PA, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (5):
  - Policlínica Privada Instituto de Medicina Nuclear, Buenos Aires, Bahia Blanca
  - Instituto Especializado Alexander Fleming, Cuidad Autónoma de Buenos Aires, Buenos Aires
  - Hospital de Gastroenterología, Loma Hermosa, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba, Córdoba Province
  - ISIS Centro Especializado, Santa Fe, Santa Fe Province
- Australia (6):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Southern Medical Day Oncology Care Centre, Wollongong, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Saint Vincent's Hospital, Fitzroy, Victoria
  - Border Medical Oncology, Murray Valley Private Hospital, Wodonga, Victoria
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Cliniques Universitaires Saint Luc, Brussels
  - Centre Hospitalier de Jolimont-Lobbes, Haine-Saint-Paul
- Brazil (9):
  - Hospital Universitario, Brasília, Federal District
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Instituto Nacional do Cancer, Rio de Janeiro, Rio de Janeiro
  - Irmandade da Santa, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - CEPON-Centro de pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital do Cancer de Barretos, Barretos, São Paulo
  - Fundacao Hospital, Jaú, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
- Cross Cancer Institute, Edmonton, Alberta, Canada
- France (7):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hôpital Saint André, Service d'Oncologie Médicale, Bordeaux
  - Clinique François Chénieux, Limoges
  - Centre Hospitalier Régional Universitaire Hôpital Saint Eloi, Montpellier
  - Centre Regional de Lutte contre le Cancer Val d'Aurelle, Montpellier
  - Centre René Gauducheau, Saint-Herblain
  - Institut Gustave-Roussy - Centre de Lutte Contre le Cancer, Villejuif
- Germany (8):
  - Ludwig-Maximilians-Universität, Medizinische Klinik und Poliklinikversität München, München, Bavaria
  - Klinikum der Ernst-Moritz-Arndt-Universität, Greifswald, Mecklenburg-Vorpommern
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Klinik der Otto-Von-Guericke-Universität Magdeburg, Magdeburg
  - Medizinische Universitätsklinik Ulm, Abt. Innere Medizin I, Ulm
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Instituto Oncologico Veneto, Oncologia Medica 1, Padua, Padova
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Ospedali Riuniti di Ancona, Torrette Di Ancona
  - Centro Ricerche Cliniche di Verona, Verona
- Vrije Universiteit Medisch Centrum, Amsterdam, North Holland, Netherlands
- Norway (2):
  - Sørlandet sykehus HF, Kristiansand
  - Oslo Universitetssykehus, Ullevål, Oslo
- Russia (13):
  - Republic Clinical Oncology Center, Izhevsk, Udmurtiya Republic
  - Regional Oncology Center, Irkutsk
  - Clinical Oncology Center #1, Krasnodar
  - Kursk Regional Oncology Center, Kursk
  - Blokhin Cancer Research Center, Moscow
  - Novosibirsk, City Clinical Hospital #1, Novosibirsk
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Mechnikov St. Petersburg State Medical Academy, Saint Petersburg
  - St. Petersburg City Oncology Center, Saint Petersburg
  - Tambov Regional Oncology Center, Tambov
  - Tula Regional Oncology Center, Tula
  - Regional Clinical Oncology Hospital, Yaroslavl
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
- Sweden (3):
  - Lanssjukhuset Ryhov, Jönköping
  - Linköping University Hospital, Linköping
  - Växjö Centrallasarettet, Vaxjo
- Ukraine (8):
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Department of Chemotherapy, Dnipropetrovsk State Medical Academy, Department of Oncology and Medical Radiology, Dnipropetrovsk
  - Public Clinical Treatment and Prophylaxis Institution "Donetsk Regional Antitumor Center", Oncosurgery Department #6, Donetsk
  - "Public Healthcare Institution ""Kharkiv Regional Clinical Oncology Center"", Abdominal Department, Kharkiv
  - National Cancer Institute, Department of Tumors of Abdominal Cavity and Retroperitoneum, Kiev
  - State Regional Diagnostics and Treatment Oncology Center, Chemotherapy Department, Lviv
  - Mykolayiv Regional Oncology Center, Surgery Department #1, Mykolayiv
  - Zakarpatya Regional Clinical Oncology Center, Chemotherapy Department, Uzhhorod
  - Clinical Facility: Public Institution "Zaporizhya City Clinical Hospital #3", Regional Center of Hepatic, Biliary Tract and Pancreatic Surgery, Surgery Department #1, Zaporizhya
- United Kingdom (3):
  - Hammersmith Hospital, London, England
  - Christie Hospital, Manchester, England
  - Beatson West of Scotland Cancer Centre, Cancer Research UK Clinical Trials Unit (CTU), Glasgow, Scotland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, multinational study conducted at 98 medical centers in Europe, Australia, and the Americas. The first patient was randomized on 04-Aug-2010 and the last patient on 09-April-2012.
Pre-assignment Details: Eligible patients were randomized (1:1) to receive either gemcitabine elaidate or gemcitabine. The stratification factors in this model were Eastern Cooperative Group Performance Status (ECOG PS) (0 vs 1) and region (North America/Western Europe/Australia vs Eastern Europe vs South America).
Groups:
- CO-1.01: CO-1.01 : 1250 mg/m2 intravenous infusion weekly for 3 weeks every 4 weeks
- Gemcitabine: Gemcitabine : 1000 mg/m2 intravenous infusion weekly for 7 weeks followed by 1 week rest, then weekly for 3 weeks every 4 weeks
Period: Overall Study
Arm/Group | CO-1.01 | Gemcitabine
Started | 182 | 185
Intent-to-Treat (ITT) Population | 182 (All randomized patients (pts)) | 185
Safety Population | 179 (All pts who received at least one dose of study drug) | 181
Tumor Evaluable Population | 178 (All pts with measurable/evaluable tumor at baseline per RECIST and have received ≥ one dose of drug) | 180
Completed | 178 | 180
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Gemcitabine Elaidate: CO-1.01 : 1250 mg/m2 intravenous infusion weekly for 3 weeks every 4 weeks
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Elaidate | Gemcitabine | Total
Number analyzed (Participants) | 182 | 185 | 367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 116 | 219
  >=65 years | 79 | 69 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.62) | 60.5 (11.19) | 61.5 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 108 | 111 | 219
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40
  Ukraine | 40 | 47 | 87
  Russian Federation | 45 | 40 | 85
  Italy | 8 | 9 | 17
  United Kingdom | 11 | 10 | 21
  France | 19 | 10 | 29
  Canada | 5 | 2 | 7
  Argentina | 2 | 6 | 8
  Brazil | 7 | 3 | 10
  Belgium | 6 | 4 | 10
  Australia | 4 | 5 | 9
  Germany | 14 | 17 | 31
  Norway | 2 | 3 | 5
  Sweden | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Patients With Low High Human Equilibrative Nucleoside Transporter 1 (hENT1) Expression
Time Frame: Monthly follow up after treatment discontinuation until death, up to 1.5 years.
Population: Analysis was per protocol and included hENT-1 low Intent to Treat (IIT) population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 114 | 118
months | 5.7 [4.7 to 7.6] | 6.1 [5.2 to 7.7]
Statistical Analysis 1: Comparison: CO-1.01 vs Gemcitabine; If the median Overall Survival (OS) for the CO-1.01-treated patients is 7.7 months and the median OS for gemcitabine-treated patients with hENT1-low status is 4 months (hazard ratio of 0.53), then a total of 144 events of death in the hENT1-low subgroup will provide over 90% power at a 0.05 (2 sided) significance level for the comparison of CO-1.01 to gemcitabine in the hENT1-low patients; Test type: Superiority or Other; p < 0.973, Log Rank; Hazard Ratio (HR) = 0.994, 95% CI 2-sided [0.746 to 1.326] — Hazard ratio and confidence interval presented above, so parameter dispersion not indicated in standard deviation field directly above

2. Secondary Outcome: Overall Survival in All Patients and Patients With hENT1 Expression
Time Frame: Monthly follow up after treatment discontinuation until death, up to 1.5 years
Population: Due to Primary endpoint showing lack of efficacy, development of CO-1.01 was stopped and secondary endpoints were not analyzed.
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: ORR, Duration of Response, and Progression Free Survival (PFS) in Patients With Measurable/Evaluable Disease, Using RECIST 1.1, up to 1.5 Years
Time Frame: Every 8 weeks
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cancer Antigen (CA)19-9 Response Rates
Time Frame: Every 4 weeks, up to 1.5 years
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Drug Tolerability and Toxicity
Time Frame: Every week, up to 1.5 years
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Pain Severity
Time Frame: Every 4 weeks, up to 1.5 years
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Health Status
Time Frame: Every 4 weeks, up to 1.5 years
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pharmacokinetic (PK) Profile of CO-1.01 Based on Sparse Sampling
Time Frame: 30 days after first dose
Population: as for outcome 2
Arm/Group | CO-1.01 | Gemcitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of informed consent to 28 days after the last study drug administration, up to 1.5 years.
Arm/Group | CO-1.01 | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 82/179 | 82/181
Other Adverse Events (participants affected / at risk) | 171/179 | 164/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CO-1.01 (N=179) | Gemcitabine (N=181)
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 2 | 0
Duodenal stenosis (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 2
Device occlusion (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 4
Cholestasis (Hepatobiliary disorders) | 2 | 6
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 2
Biliary sepsis (Infections and infestations) | 1 | 4
Biliary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 1 | 2
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneuomococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Pneuomothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 5
C-reactive protein increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 39
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Couth (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Arterial thrombosis limb (Vascular disorders) | 9 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 3 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Obstruction gastric (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 2 | 1
Infection (not confirmed) due to fever and elevated CRP (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CO-1.01 (N=179) | Gemcitabine (N=181)
Nausea (Gastrointestinal disorders) | 70 | 59
Anaemia (Blood and lymphatic system disorders) | 65 | 78
Thrombocytopenia (Blood and lymphatic system disorders) | 53 | 60
Asthenia (General disorders) | 47 | 34
Neutropenia (Blood and lymphatic system disorders) | 46 | 47
Decreased appetite (Gastrointestinal disorders) | 42 | 33
Vomiting (Gastrointestinal disorders) | 41 | 35
Fatigue (General disorders) | 38 | 45
Pyrexia (General disorders) | 35 | 41
Diarrhoea (Gastrointestinal disorders) | 34 | 30
Abdominal pain (Gastrointestinal disorders) | 32 | 24
Constipation (Gastrointestinal disorders) | 26 | 25
Oedema peripheral (General disorders) | 25 | 34
Alanine aminotransferase increased (Investigations) | 20 | 15
Abdominal pain upper (Gastrointestinal disorders) | 19 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 24
Aspartate aminotransferase increased (Investigations) | 16 | 19
Platelet count decreased (Blood and lymphatic system disorders) | 14 | 10
Weight decreased (Investigations) | 14 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 16
Insomnia (Psychiatric disorders) | 13 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Leukopenia (Blood and lymphatic system disorders) | 12 | 17
Blood akaline phosphatase increased (Investigations) | 11 | 10
Dizziness (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 11 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 11 | 17
Thrombocytosis (Blood and lymphatic system disorders) | 10 | 1
Gamma-glutamyltransferase increased (Investigations) | 9 | 8
Ascites (Gastrointestinal disorders) | 7 | 17
Hypertension (Vascular disorders) | 7 | 10
Hypotension (Vascular disorders) | 5 | 10
Urinary tract infection (Infections and infestations) | 5 | 11

LIMITATIONS AND CAVEATS:
Due to Primary endpoint showing lack of efficacy, development of CO-1.01 was stopped and secondary endpoints were not analyzed. However, patient enrollment completed normally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.